CLINICAL TRIAL: NCT00633035
Title: Comparison of Esomeprazole and Famotidine for Stress Ulcer Prophylaxis in Neurosurgical Intensive Care Unit
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tzong-Hsi Lee, Chief of Division of Hepatology and Gastroenterology, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FEMH-94-C-016
Record Dates: First submitted 2008-03-03; First posted 2008-03-11 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Ulcer
Keywords: ulcer; esomeprazole; famotidine; Neurosurgery
MeSH Terms: conditions — Ulcer | interventions — Esomeprazole; Famotidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): oral esomeprazole tablet dissolved in water given through NG tube
  Interventions: Drug: esomeprazole 40 mg
- 2 (Active Comparator): intravenous famotidine injection
  Interventions: Drug: famotidine 20 mg

INTERVENTIONS:
Drug: esomeprazole 40 mg — esomeprazole 40 mg po given for 7 days
  Other Names: Nexium
  Arms: 1
Drug: famotidine 20 mg — famotidine 20 mg intravenous bolus q12h for 7 days
  Other Names: gaster
  Arms: 2

SUMMARY:
Although stress ulcer is a complication that can cause mortality and morbidity in critical patients, there is still lack of consensus about its prophylaxis. There is also few data available from Taiwan. H2 blockers are commonly used due to convenience. Some prefer sucralfate (a mucosal protective agent) for the sake of less associated nosocomial pneumonia. Recently, proton pump inhibitors were shown to have good prophylactic effects for stress ulcer. Esomeprazole, an isoform of omeprazole, has good acid suppression effect and the tablets are soluble for the use of tube feeding. Our previous study showed that there was no difference for the efficacy of stress ulcer prophylaxis between esomeprazole and sucralfate in patients admitted to medical ICU with at least one risk factor. The prevalence of nosocomial pneumonia was also similar.

We will enroll those patients that have received intracranial surgery and admitted to neurosurgical ICU. After obtaining the consent, we will give them prophylactic drugs for 7 days within 24 hours. They are randomly allocated to 2 groups. Group I: esomeprazole 40 mg qd from NG route or orally; Group II: famotidine 20 mg iv bolus q12h. We will monitor the following data: Glasgow coma scale, APACHE II score, CBC, CXR, stool character and OB test, NG aspirate. If clinical evidence of UGI bleeding occurs, endoscopy will be performed. We define the end point as overt bleeding, death or transfer out of ICU. We will compare the prevalence of UGI bleeding and nosocomial pneumonia in these 2 groups.

DETAILED DESCRIPTION:
1. patients: the patients receiving neurosurgery and admitted to intensiv care unit within 24 hours. They are enrolled after well explanation and giving written consdent. Those are less than 18 y/o, pregnant, not suitable for NG feeding, already having GI bleeding, are excluded
2. grouping & intervention: The patients are randomized to 2 groups. 1st group:receiving esomeprazole 40 mg qd via NG; 2nd group: receiving famotidine 20 mg iv bolus q12h. These medication are used for 7 days. Estimated enrolled number is 60 for each group
3. monitoring: Glasgow coma scale , APACHE II score at baseline, CBC、CXR at basleine and qod, stool OB q3d，NG drainage、sputum、 stool character, ICU routine （TPR, BP）, ICU admitted day, 30 day mortality rate. UGI endoscopy arranged according judgement of attending doctors
4. end points: overt UGI bleeding（tarry stool,hematemesis、coffee ground substance from NG more than 60 ml, Hb decrease more than 2g/dl and endoscopic proof of bleeder）. ventilator associated pneumonia: new onset and persisted hazziness in CXR, combined with fever, leucocytosis and positive sputum smear finding.
5. statistics: the prevalence of overt bleeding and ventilator associated pneumonia is examined by Fisher's exact test, the demongraphic data and disease severity data are examined by student's t test or Chi-square test。

ELIGIBILITY:
Inclusion Criteria:

* Within 24 hours of admission to Neurosurgical ICU after neurosurgery with ventilator support

Exclusion Criteria:

* Less than 18 y/o;
* Pregnancy;
* Not suitable for medication from NG route,
* Had GI bleeding at admission to ICU

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-09; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
UGI bleeding: hematemesis or much coffee ground substance (> 60 ml) from NG, tarry stool, decrease of Hb more than 2g/dl and endoscopic proof of bleeder | 7 days within the period of prophylactic medication use

SECONDARY OUTCOMES:
ventilator associated pneumonia: new onset and persistent hazziness in CXR 48 hours after admission to ICU, combined with fever and leucocytosis and positive sputum smear finding | 7 days within the period of prophyactic medication use

CONTACTS AND LOCATIONS:
Overall Officials: Tzong-Hsi Lee, M.D., Principal Investigator — Far Eastern Memorial Hospital, Taipei, Taiwan
Locations (1):
- Far Eastern Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Cook DJ, Fuller HD, Guyatt GH, Marshall JC, Leasa D, Hall R, Winton TL, Rutledge F, Todd TJ, Roy P, et al. Risk factors for gastrointestinal bleeding in critically ill patients. Canadian Critical Care Trials Group. N Engl J Med. 1994 Feb 10;330(6):377-81. doi: 10.1056/NEJM199402103300601. PMID 8284001
- [Background] Maier RV, Mitchell D, Gentilello L. Optimal therapy for stress gastritis. Ann Surg. 1994 Sep;220(3):353-60; discussion 360-3. doi: 10.1097/00000658-199409000-00011. PMID 8092901
- [Background] Lam NP, Le PD, Crawford SY, Patel S. National survey of stress ulcer prophylaxis. Crit Care Med. 1999 Jan;27(1):98-103. doi: 10.1097/00003246-199901000-00034. PMID 9934901
- [Background] Cook DJ, Reeve BK, Guyatt GH, Heyland DK, Griffith LE, Buckingham L, Tryba M. Stress ulcer prophylaxis in critically ill patients. Resolving discordant meta-analyses. JAMA. 1996 Jan 24-31;275(4):308-14. PMID 8544272
- [Background] Allen ME, Kopp BJ, Erstad BL. Stress ulcer prophylaxis in the postoperative period. Am J Health Syst Pharm. 2004 Mar 15;61(6):588-96. doi: 10.1093/ajhp/61.6.588. PMID 15061430
- [Background] Kantorova I, Svoboda P, Scheer P, Doubek J, Rehorkova D, Bosakova H, Ochmann J. Stress ulcer prophylaxis in critically ill patients: a randomized controlled trial. Hepatogastroenterology. 2004 May-Jun;51(57):757-61. PMID 15143910
- [Background] Tryba M, Cook D. Current guidelines on stress ulcer prophylaxis. Drugs. 1997 Oct;54(4):581-96. doi: 10.2165/00003495-199754040-00005. PMID 9339962
- [Background] Driks MR, Craven DE, Celli BR, Manning M, Burke RA, Garvin GM, Kunches LM, Farber HW, Wedel SA, McCabe WR. Nosocomial pneumonia in intubated patients given sucralfate as compared with antacids or histamine type 2 blockers. The role of gastric colonization. N Engl J Med. 1987 Nov 26;317(22):1376-82. doi: 10.1056/NEJM198711263172204. PMID 2891032
- [Background] Fabian TC, Boucher BA, Croce MA, Kuhl DA, Janning SW, Coffey BC, Kudsk KA. Pneumonia and stress ulceration in severely injured patients. A prospective evaluation of the effects of stress ulcer prophylaxis. Arch Surg. 1993 Feb;128(2):185-91; discussion 191-2. doi: 10.1001/archsurg.1993.01420140062010. PMID 8431119
- [Background] Levy MJ, Seelig CB, Robinson NJ, Ranney JE. Comparison of omeprazole and ranitidine for stress ulcer prophylaxis. Dig Dis Sci. 1997 Jun;42(6):1255-9. doi: 10.1023/a:1018810325370. PMID 9201091
- [Background] Lasky MR, Metzler MH, Phillips JO. A prospective study of omeprazole suspension to prevent clinically significant gastrointestinal bleeding from stress ulcers in mechanically ventilated trauma patients. J Trauma. 1998 Mar;44(3):527-33. doi: 10.1097/00005373-199803000-00020. PMID 9529184
- [Background] Daley RJ, Rebuck JA, Welage LS, Rogers FB. Prevention of stress ulceration: current trends in critical care. Crit Care Med. 2004 Oct;32(10):2008-13. doi: 10.1097/01.ccm.0000142398.73762.20. PMID 15483408
- [Background] Lu WY, Rhoney DH, Boling WB, Johnson JD, Smith TC. A review of stress ulcer prophylaxis in the neurosurgical intensive care unit. Neurosurgery. 1997 Aug;41(2):416-25; discussion 425-6. doi: 10.1097/00006123-199708000-00017. PMID 9257310
- [Background] Martin LF, Booth FV, Karlstadt RG, Silverstein JH, Jacobs DM, Hampsey J, Bowman SC, D'Ambrosio CA, Rockhold FW. Continuous intravenous cimetidine decreases stress-related upper gastrointestinal hemorrhage without promoting pneumonia. Crit Care Med. 1993 Jan;21(1):19-30. doi: 10.1097/00003246-199301000-00009. PMID 8420726
- [Background] Hatton J, Lu WY, Rhoney DH, Tibbs PA, Dempsey RJ, Young B. A step-wise protocol for stress ulcer prophylaxis in the neurosurgical intensive care unit. Surg Neurol. 1996 Nov;46(5):493-9. doi: 10.1016/s0090-3019(96)00245-5. PMID 8874553